CLINICAL TRIAL: NCT06380439
Title: The Effect of Wrist Ankle Acupuncture on Post-Total Hip Arthroplasty Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Wijayani Mardiana, medical doctore, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-10-1763
Record Dates: First submitted 2024-04-08; First posted 2024-04-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Hip Osteoarthritis; Hip Fractures; Hip Injuries
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Hip; Hip Fractures; Hip Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wrist ankle acupuncture (Experimental): wrist ankle acupuncture using 0.25 x 25mm filiform needle on lower 1, lower 4, lower 5 area ipsilateral to the surgical side, then covered with 5cm long micropore, retention for 4 hours
  Interventions: Procedure: wrist ankle acupuncture
- sham wrist ankle acupuncture (Sham Comparator): 0.25 x 25mm filiform needle pricked and placed on the surface of the skin on lower 1, lower 4, lower 5 area ipsilateral to the surgical side, covered with 5cm long micropore, retention for 4 hours
  Interventions: Procedure: wrist ankle acupuncture

INTERVENTIONS:
Procedure: wrist ankle acupuncture — wrist ankle acupuncture: wrist ankle acupuncture using 0.25 x 25mm filiform needle on lower 1, lower 4, lower 5 area ipsilateral to the surgical side, then covered with 5cm long micropore, retention for 4 hours

SUMMARY:
Total hip arthroplasty is one of the most cost-effective orthopedic surgical procedures which can restore hip function and improve the patient's quality of life. However, total hip arthroplasty is significantly associated with postoperative pain. Pain after total hip arthroplasty surgery can adversely affect the patient's early postoperative recovery, postoperative mobility, and hinder rehabilitation.

Wrist ankle acupuncture (WAA) is a simpler acupuncture technique, using fewer points, shallow needle insertion and lighter stimulation. Wrist-ankle acupuncture as multimodal analgesia after orthopedic surgery is useful for reducing pain and reduce the incidence of post-surgical side effects. The primary aim of this study is to investigate whether wrist ankle acupuncture therapy gives better and results for post total hip arthroplasty pain than sham wrist ankle acupuncture

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate and compare the effects of wrist ankle acupuncture and sham wrist ankle acupuncture as a therapy for post total hip arthroplasty pain. The subjects are 32 males/female who just undergone total hip arthroplasty surgery and has returned to inpatient ward. They will be randomly assigned to 2 groups: (1) wrist ankle acupuncture and (2) Sham wrist ankle acupuncture. The subjects will receive two sessions of treatment. The outcome will be assessed before treatment (baseline), after fist acupuncture session, after second acupuncture session and a day after the second session. Patients and the outcome assessors will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective primary total hip arthroplasty surgery at dr. Cipto Mangunkusumo Hospital, Persahabatan Hospital, andFatmawati Hospital
2. Aged over 18 years
3. Willing to sign informed consent

Exclusion Criteria:

1. Have a history of malignancy
2. Revision total hip arthroplasty patient
3. Post-total hip surgery patient treated in ICU.
4. The patient has a mental disorder so he cannot understand the explanation given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | after the surgery when the patient has returned to the inpatient ward (before the 1st acupuncture session), 4 hours since the 1st measure (after 1st acupuncture session), one day after the 1st measure (after 2nd acupuncture), 2 days after 1st measure
  Pain rating scale for measuring pain

SECONDARY OUTCOMES:
recovery rate | monitored since day 1 after surgery up to 4 days
  the time when patient starts to learn to walk with assistive device

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - RSCM
Locations (3):
- Indonesia (3):
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region
  - Fatmawati Hospital, Jakarta
  - Persahabatan Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No